CLINICAL TRIAL: NCT04606784
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Nebulized Ampion In Adults With Respiratory Distress Secondary to COVID-19 Infection
Brief Title: Study of Nebulized Ampion for the Treatment of Adult COVID-19 Patients With Respiratory Distress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP-014
Record Dates: First submitted 2020-10-27; First posted 2020-10-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — aspartyl-alanyl-diketopiperazine; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ampion (Experimental): Ampion
  Interventions: Biological: Ampion; Other: Standard of Care
- Standard of Care (Other): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Ampion — Ampion, nebulized for inhalation
  Arms: Ampion
Other: Standard of Care — Standard of Care

SUMMARY:
This is a Phase 1 randomized study to evaluate the safety, tolerability and efficacy of nebulized Ampion in improving the clinical course and outcomes of patients hospitalized with COVID-19 infection who have respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years old.
2. Diagnosed with COVID-19, as evaluated by PCR test confirming infection with SARS-CoV-2, or suspected COVID-19 diagnosis based on radiological clinical findings.
3. Respiratory distress as evidenced by at least two of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.)
   * Recording of SpO2 ≤ 90% or the patient is requiring supplemental oxygen to maintain an SpO2 ≥ 90%
   * Requiring supplemental oxygen
   * Diagnosis of mild, moderate, or severe ARDS by Berlin definition
4. A signed informed consent form from the patient or the patient's legal representative must be available.

Exclusion Criteria:

1. In the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
2. Patient has a do-not-resuscitate (DNR) or do-not-intubate (DNI) order in place
3. Patient has severe chronic obstructive pulmonary disease (COPD), chronic renal failure, or significant liver abnormality (e.g. cirrhosis, transplant, etc.).
4. Patient is on chronic immunosuppressive medication.
5. As a result of the medical review and screening investigation, the Principal Investigator considers the patient unfit for the study.
6. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion) or excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
7. Patient has known pregnancy or is currently breastfeeding.
8. Participation in another clinical trial (not including treatments for COVID-19 as approved by the FDA through expanded access or compassionate use).
9. Baseline QT prolongation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Day 5
  Incidence and severity of adverse events
Incidence and severity of adverse events | Day 28
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Clinical status using 8-point ordinal scale | Day 5
  Efficacy measures for clinical improvement using 8-point ordinal scale: 0 = Uninfected, 1 = Ambulatory without limitation of activity, 2 = Ambulatory with limitation of activity, 3 = Hospitalized mild disease, no oxygen, 4 = Hospitalized mild disease, supplemental oxygen, 5 = Hospitalized severe disease, non-invasive ventilation or high-flow oxygen, 6 = Hospitalized severe disease, intubation and mechanical ventilation, 7 = Hospitalized severe disease, ventilation plus additional organ support, 8 = Death
Clinical status using 8-point ordinal scale | Day 28
  Efficacy measures for clinical improvement using 8-point ordinal scale: 0 = Uninfected, 1 = Ambulatory without limitation of activity, 2 = Ambulatory with limitation of activity, 3 = Hospitalized mild disease, no oxygen, 4 = Hospitalized mild disease, supplemental oxygen, 5 = Hospitalized severe disease, non-invasive ventilation or high-flow oxygen, 6 = Hospitalized severe disease, intubation and mechanical ventilation, 7 = Hospitalized severe disease, ventilation plus additional organ support, 8 = Death

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Colorado Springs, Colorado, United States

REFERENCES:
- [Derived] Roshon M, Lemos-Filho L, Cherevka H, Goldberg L, Salottolo K, Bar-Or D. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of a Novel Inhaled Biologic Therapeutic in Adults with Respiratory Distress Secondary to COVID-19 Infection. Infect Dis Ther. 2022 Feb;11(1):595-605. doi: 10.1007/s40121-021-00562-z. Epub 2021 Nov 14. PMID 34775578